CLINICAL TRIAL: NCT00024167
Title: A Prospective Randomized Phase III, Trial Comparing Consolidation Therapy With or Without Strontium-89 Following Induction Chemotherapy in Androgen-Independent Prostate Cancer
Brief Title: Chemotherapy With or Without Strontium-89 in Treating Patients With Prostate Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated due to slow accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID00-156; U10CA045809 (NIH); P30CA016672 (NIH); MDA-ID-00156 (Other: UT MD Anderson Cancer Center); NCI-3410; CDR0000068897 (Registry Identifier: NCI PDQ); NCI-2009-00009 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Results first posted 2016-03-22 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-02

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IV prostate cancer; recurrent prostate cancer; Strontium-89; Induction Chemotherapy; Androgen-Independent Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Doxorubicin; Estramustine; Ketoconazole; Prednisone; Vinblastine; strontium chloride; Strontium-89; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Induction regimen A (Experimental): Doxorubicin IV over 24 hours day 1; Oral ketoconazole 3 x daily on days 1-7 of weeks 1, 3, and 5; Vinblastine IV over 30 minutes Day 1, oral Estramustine 3 x daily on Days 1-7 of weeks 2, 4, and 6.
  Interventions: Drug: Doxorubicin hydrochloride; Drug: Estramustine phosphate sodium; Drug: Ketoconazole; Drug: Vinblastine
- Induction regimen B (Experimental): Oral Prednisone 2 x daily on days 1-21 (days 1-14 of course 5 only) and Docetaxel IV over 1 hour Day 1.
  Interventions: Drug: Docetaxel; Drug: Prednisone; Drug: Dexamethasone
- Consolidation arm I (Experimental): Doxorubicin IV over 24 hours once weekly for 6 weeks + Strontium-89 IV once at beginning of chemotherapy.
  Interventions: Drug: Doxorubicin hydrochloride; Radiation: Strontium chloride Sr 89
- Consolidation arm II (Experimental): Doxorubicin as in Consolidation arm I.
  Interventions: Drug: Doxorubicin hydrochloride

INTERVENTIONS:
Drug: Docetaxel — 75 mg/m2 intravenous piggyback (IVPB) over 1 hour, Day 1, every 3 weeks.
  Other Names: Taxotere
  Arms: Induction regimen B
Drug: Doxorubicin hydrochloride — 20 mg/m2 IV, day 1 on Weeks 1, 3, 5
  Other Names: Adriamycin PFS; Adriamycin RDF; Doxorubicin
  Arms: Consolidation arm I; Consolidation arm II; Induction regimen A
Drug: Estramustine phosphate sodium — 140 mg orally 3 x day, Days 1 through 7 on Weeks 2, 4, 6
  Other Names: Estramustine
  Arms: Induction regimen A
Drug: Ketoconazole — 400 mg orally (po) 3 x day, Days 1 through 7
  Other Names: Nizoral
  Arms: Induction regimen A
Drug: Prednisone — 5 mg orally 2 x daily, weeks 1-14
  Arms: Induction regimen B
Drug: Vinblastine — 4 mg/m2 IVPB, Day 1 on Weeks 2, 4, 6
  Other Names: Velban
  Arms: Induction regimen A
Radiation: Strontium chloride Sr 89 — One dose (4 mCi total dose) IV
  Other Names: strontium-89 chloride; Sr-89; strontium-89; Metastron
  Arms: Consolidation arm I
Drug: Dexamethasone — 4 mg is given orally at 12 and 1 hours before and 12 hours after docetaxel.
  Other Names: Decadron
  Arms: Induction regimen B

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radioactive substances such as strontium-89 may relieve bone pain associated with prostate cancer. It is not yet known whether chemotherapy is more effective with or without strontium-89 in treating bone metastases.

PURPOSE: This randomized phase III trial is studying giving chemotherapy together with strontium-89 to see how well it works compared to chemotherapy alone in treating patients with prostate cancer that has spread to the bone.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effectiveness, in terms of overall survival, of consolidation therapy with or without strontium chloride Sr 89 after induction chemotherapy in patients with androgen-independent prostate cancer.

OUTLINE: This is a randomized study. Patients are stratified according to type of induction chemotherapy (KAVE vs prednisone and docetaxel), number of bony metastases (no more than 20 vs more than 20), Eastern Cooperative Oncology (ECOG) performance status (0-1 vs 2-3), and use of zoledronate (yes vs no).

* Induction therapy: Patients receive 1 of 2 induction therapy regimens.

  * Regimen A (KAVE): Patients receive doxorubicin IV over 24 hours on day 1 and oral ketoconazole three times daily on days 1-7 of weeks 1, 3, and 5. Patients receive vinblastine IV over 30 minutes on day 1 and oral estramustine three times daily on days 1-7 of weeks 2, 4, and 6. Patients receive no treatment on weeks 7 and 8. Treatment repeats every 8 weeks for at least 2 courses* in the absence of disease progression or unacceptable toxicity.

NOTE: *Patients continue to receive oral ketoconazole three times daily until disease progression.

* Regimen B (prednisone and docetaxel): Patients receive oral prednisone twice daily on days 1-21 (days 1-14 of course 5 only) and docetaxel IV over 1 hour on day 1. Treatment repeats every 21 days for at least 5 courses in the absence of disease progression or unacceptable toxicity.

  * Consolidation therapy: Patients with a prostate-specific antigen (PSA) response (at least 50% decline in PSA level from baseline at week 16 OR at least 2 PSA levels decreased at least 50% from baseline) are randomized to 1 of 2 consolidation treatment arms.
* Arm I: Patients receive doxorubicin IV over 24 hours once weekly for 6 weeks plus strontium chloride Sr 89 IV once at the beginning of chemotherapy.
* Arm II: Patients receive doxorubicin as in arm I. Patients are followed every 4 weeks until PSA progression and then every 3 months thereafter.

PROJECTED ACCRUAL: Approximately 480 patients (240 randomized) will be accrued for this study within 48 months.

ELIGIBILITY:
Inclusion Criteria:

1. Rising PSA on at least 2 occasions >1 week apart (minimum value of 5 ng/ml), accompanied either by bone pain or, if the patient is asymptomatic, by a worsening bone scan with new lesions over a period of <6 months
2. Patients on antiandrogens should be discontinued from flutamide or nilutamide for at least 4 weeks and bicalutamide for 6 weeks; If progression is documented during this time interval as in inclusion criterion # 1, patients are eligible
3. Osteoblastic metastases on bone scan or CT scan
4. Androgen-independent prostate adenocarcinoma
5. Castrate testosterone level </= 50 ng/ml; treatment to maintain castrate levels of testosterone must be continued
6. >/= 18 years of age
7. Life expectancy of greater than or equal to 12 weeks
8. Zubrod performance status </= 3
9. Patients must have normal organ and marrow function as defined below: Leukocytes greater than 3,000/mcL Absolute neutrophil count greater than 1,500/mcL Platelets greater than 100,000/mcL Total bilirubin less than or equal to 2X institutional upper limit of normal AST(SGOT)/ALT(SGPT) less than or equal to 2X institutional upper limit of normal
10. The patient must have the ability to understand and the willingness to sign a written informed consent document
11. Participating subjects and their female partners agree to the use of adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation

Exclusion Criteria:

1. History of allergic reactions attributed to compounds of similar chemical or biologic composition to the agents used on this trial
2. Prior doxorubicin, or vinblastine in the KAVE arm and prior docetaxel in the prednisone plus docetaxel arm. However, previous treatment using other secondary hormonal agents (aminoglutethimide, diethylstilbesterol, estramustine), steroids (dexamethasone, prednisone, hydrocortisone), angiogenesis inhibitors, gene therapy, or immunotherapy are allowed
3. More than one prior cytotoxic treatment
4. Prior Sr-89 or Sm-153 treatment
5. Patients who have had chemotherapy, immunotherapy, or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
6. Previous vagotomy or other conditions (such as pernicious anemia) associated with achlorhydria. Patients with active peptic ulcer disease who still require regular use of H2 blockers (such as cimetidine [Tagamet], ranitidine [Zantac], famotidine [Pepcid], etc), proton pump inhibitors (omeprazole [Prilosec]), or antacids (Mylanta, Maalox, Tums, etc) at week 16 of induction chemotherapy (option 1 only) might not be suitable for randomization
7. Predominant visceral metastases in the liver, lungs, or brain
8. Symptomatic lymphadenopathy (scrotal or pedal edema) or significant local invasive disease (hematuria)
9. Small cell carcinoma
10. Recent history of transient ischemic attacks (TIA) or myocardial infarctions (MI) within 12 months, or active angina or claudication sufficient to limit activity
11. Active or likely to become active second malignancy (other than non-melanoma skin cancer)
12. Uncontrolled inter-current illness: including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2002-04; Primary Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shi-Ming Tu, MD, Study Chair — M.D. Anderson Cancer Center
Locations (40):
- United States (40):
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Veterans Affairs Medical Center - Hines, Hines, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Kinston Medical Specialists, Kinston, North Carolina
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Barberton Citizens Hospital, Barberton, Ohio
  - Cancer Care Center, Incorporated, Salem, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - McLeod Regional Medical Center, Florence, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Medical City Dallas Hospital, Dallas, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Result] Tu SM, Kim J, Pagliaro LC, Vakar-Lopez F, Wong FC, Wen S, General R, Podoloff DA, Lin SH, Logothetis CJ. Therapy tolerance in selected patients with androgen-independent prostate cancer following strontium-89 combined with chemotherapy. J Clin Oncol. 2005 Nov 1;23(31):7904-10. doi: 10.1200/JCO.2005.01.2310. PMID 16258090
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: April 16, 2002 to October 20, 2010 from various hospitals and institutions representing the Community Clinical Oncology Program (CCOP).
Pre-assignment Details: Of the 265 participants enrolled - 127 were randomized to either the Sr-89 treatment arm or the no Sr-89 treatment arm and the rest (138 participants) did not qualify for randomization. Of the 138 participants, 5 did not receive any treatment and the rest received only induction treatment. Study was closed prematurely due to issues with accrual.
Groups:
- Induction Treatment + Strontium-89: Induction treatment option 1: Weeks 1,3,5: Doxorubicin 20 mg/m^2 IV, day 1 and Ketoconazole 400 mg oral 3 x daily, days 1 through 7. Weeks 2,4,6: Vinblastine 4 mg/m^2 IVPB, day 1 and Estramustine 140 mg oral 3 x daily, days 1 through 7. Weeks 7,8: No treatment. Hydrocortisone 10 mg oral 2 x daily will be administered throughout treatment or Induction treatment option 2: Prednisone 5 mg oral 2 x daily, weeks 1-14 and Docetaxel 75 mg/m^2 IVPB over 1 hour, every 3 weeks. Dexamethasone 4 mg is given orally at 12 and 1 hours before and 12 hours after docetaxel. Randomization: Doxorubicin IV over 24 hours once weekly for 6 weeks + Strontium-89 IV once at beginning of chemotherapy.
- Induction Treatment + No Strontium-89: Induction treatment option 1: Weeks 1,3,5: Doxorubicin 20 mg/m^2 IV, day 1 and Ketoconazole 400 mg oral 3 x daily, days 1 through 7. Weeks 2,4,6: Vinblastine 4 mg/m^2 IVPB, day 1 and Estramustine 140 mg oral 3 x daily, days 1 through 7. Weeks 7,8: No treatment. Hydrocortisone 10 mg oral 2 x daily will be administered throughout treatment or Induction treatment option 2: Prednisone 5 mg oral 2 x daily, weeks 1-14 and Docetaxel 75 mg/m^2 IVPB over 1 hour, every 3 weeks. Dexamethasone 4 mg is given orally at 12 and 1 hours before and 12 hours after docetaxel. Randomization: Doxorubicin 20mg/m^2 IV over 24 hours once weekly for 6 weeks.
Period: Overall Study
Arm/Group | Induction Treatment + Strontium-89 | Induction Treatment + No Strontium-89
Started | 65 | 62
Induction Treatment Option 1 Completed | 22 | 21
Induction Treatment Option 2 Completed | 43 | 41
Completed | 12 | 15
Not Completed | 53 | 47
Not completed — Death | 53 | 47

BASELINE CHARACTERISTICS:
Population: Of the 265 participants enrolled - 133 participants received only induction treatment and 127 were randomized to either the Sr-89 treatment arm or the no Sr-89 treatment arm. 5 participants never received any treatment.
Groups:
- Induction Treatment: Induction treatment option 1: Weeks 1,3,5: Doxorubicin 20 mg/m^2 IV, day 1 and Ketoconazole 400 mg oral 3 x daily, days 1 through 7. Weeks 2,4,6: Vinblastine 4 mg/m^2 IVPB, day 1 and Estramustine 140 mg oral 3 x daily, days 1 through 7. Weeks 7,8: No treatment. Hydrocortisone 10 mg oral 2 x daily will be administered throughout treatment or Induction treatment option 2: Prednisone 5 mg oral 2 x daily, weeks 1-14 and Docetaxel 75 mg/m^2 IVPB over 1 hour, every 3 weeks. Dexamethasone 4 mg is given orally at 12 and 1 hours before and 12 hours after docetaxel.
- Total: Total of all reporting groups
Arm/Group | Induction Treatment | Induction Treatment + Strontium-89 | Induction Treatment + No Strontium-89 | Total
Number analyzed (Participants) | 133 | 65 | 62 | 260
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 1 | 1
  Between 18 and 65 years | 53 | 22 | 23 | 98
  >=65 years | 80 | 43 | 38 | 161
Age, Continuous [Median (Full Range); unit: years] | 67 [44 to 85] | 68 [48 to 85] | 67 [8 to 80] | 67 [8 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 133 | 65 | 62 | 260
Region of Enrollment [Number; unit: participants]
  United States | 133 | 65 | 62 | 260

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival From Randomization
Description: Overall survival (OS) was computed using the number of months from the date of randomization to the date of death. Participants still alive were censored at the last follow-up date. Kaplan-Meier methodology was used to evaluate OS.
Time Frame: Followed every 4 weeks from randomization until death, up to 7 years.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Induction Treatment + Strontium-89: Induction treatment option 1 or induction treatment option 2. Randomization: Doxorubicin IV over 24 hours once weekly for 6 weeks + Strontium-89 IV once at beginning of chemotherapy.
- Induction Treatment + No Strontium-89: Induction treatment option 1 or induction treatment option 2. Randomization: Doxorubicin 20mg/m^2 IV over 24 hours once weekly for 6 weeks.
Arm/Group | Induction Treatment + Strontium-89 | Induction Treatment + No Strontium-89
Number analyzed (Participants) | 65 | 62
months | 24.2 [19.8 to 29.8] | 22.8 [17.7 to 27.7]

2. Secondary Outcome: Overall Survival From Registration
Description: Overall survival (OS) was computed using the number of months from the date of registration to the date of death. Participants still alive were censored at the last follow-up date. Kaplan-Meier methodology was used to evaluate OS.
Time Frame: Followed every 4 weeks from registration until death, up to 7 years.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Induction Treatment + Strontium-89 | Induction Treatment + No Strontium-89
Number analyzed (Participants) | 65 | 62
months | 27.9 [23.6 to 34.2] | 26.6 [21.1 to 32.2]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious adverse events (SAEs) were collected from administration of induction therapy to discontinuation of study drug. Overall collection period: June 2002 to July 2014.
Groups:
- Induction Treatment: Induction treatment option 1 or induction treatment option 2.
Arm/Group | Induction Treatment | Induction Treatment + Strontium-89 | Induction Treatment + No Strontium-89
Serious Adverse Events (participants affected / at risk) | 77/138 | 53/65 | 47/62
Other Adverse Events (participants affected / at risk) | 34/138 | 12/65 | 13/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction Treatment (N=138) | Induction Treatment + Strontium-89 (N=65) | Induction Treatment + No Strontium-89 (N=62)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Infection with Grade 3 or 4 Neutrophils (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Spinal Cord Compression (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 77 (77) | 53 (53) | 47 (47)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neutrophil Count Decreased (Blood and lymphatic system disorders) | 1 (1) | 4 (4) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0)
Hemoglobin Decreased (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0)
Blood Glucose Increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 1 (1) | 0 (0)
Lymphopenia (Infections and infestations) | 2 (3) | 1 (3) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 2 (2) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Peripheral Motor Neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Serum Phosphate Decreased (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Aspartate Aminotransferase Increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Serum Sodium Decreased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Psychosis (Psychiatric disorders) | 1 (2) | 0 (0) | 0 (0)
Anxiety (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Alkaline Phosphatase Increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Constitutional Symptoms (General disorders) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction Treatment (N=138) | Induction Treatment + Strontium-89 (N=65) | Induction Treatment + No Strontium-89 (N=62)
Bone Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 2 (2)
Nausea (Gastrointestinal disorders) | 11 (14) | 2 (2) | 5 (7)
Vomiting (Gastrointestinal disorders) | 7 (9) | 0 (0) | 1 (1)
Fatigue (General disorders) | 16 (18) | 11 (16) | 5 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 2 (2) | 3 (3)
Edema Limbs (Blood and lymphatic system disorders) | 8 (10) | 5 (6) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Metabolism and nutrition disorders) | 1 (1) | 1 (4) | 1 (1)
Bilirubin Increased (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Aspartate Aminotransferase Increased (Metabolism and nutrition disorders) | 5 (5) | 1 (2) | 1 (1)
Neutrophil Count Decreased (Blood and lymphatic system disorders) | 1 (2) | 1 (2) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (3) | 3 (4)
Platelet Count Decreased (Blood and lymphatic system disorders) | 2 (3) | 2 (2) | 1 (1)
Mucositis Oral (Gastrointestinal disorders) | 1 (2) | 2 (3) | 1 (1)
Serum Potassium Decreased (Metabolism and nutrition disorders) | 2 (2) | 1 (3) | 2 (2)
Alkaline Phosphatase Increased (Metabolism and nutrition disorders) | 3 (6) | 1 (1) | 2 (2)
Anorexia (Gastrointestinal disorders) | 6 (7) | 1 (1) | 1 (1)
Insomnia (General disorders) | 5 (5) | 1 (1) | 1 (1)
Blood Glucose Increased (Metabolism and nutrition disorders) | 6 (7) | 1 (3) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 2 (2) | 1 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (3) | 0 (0)
Serum Sodium Decreased (Metabolism and nutrition disorders) | 2 (3) | 3 (8) | 0 (0)
Neurology (Other) (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Urinary Frequency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 2 (2)
Peripheral Sensory Neuropathy (Nervous system disorders) | 8 (8) | 2 (2) | 1 (1)
Blood/Bone Marrow (Other) (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Serum Cacium Decreased (Metabolism and nutrition disorders) | 4 (8) | 1 (7) | 1 (1)
Lymphopenia (Blood and lymphatic system disorders) | 2 (5) | 1 (10) | 1 (1)
Hypersensitivity (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Rash Acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Nail Disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 10 (10) | 3 (4) | 2 (2)
Serum Albumin Decreased (Metabolism and nutrition disorders) | 4 (10) | 1 (4) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 1 (4) | 2 (7) | 1 (2)
Creatinine Increased (Metabolism and nutrition disorders) | 1 (1) | 1 (4) | 0 (0)
Hypotension (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Infection (Other) (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Peripheral Motor Neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Metabolic/Laboratory (Other) (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal (Other) (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
INR Increased (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Watering Eyes (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Taste Alteration (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Hot Flashes (Endocrine disorders) | 3 (3) | 1 (1) | 0 (0)
Anxiety (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Auditory/Ear (Other) (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constitutional Symptoms (Other) (General disorders) | 1 (1) | 1 (1) | 0 (0)
Blood Uric Acid Increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatology/Skin (Other) (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Dry Mouth (General disorders) | 0 (0) | 1 (1) | 1 (1)
Renal/Genitourinary (Other) (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Erectile Dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Libido Decreased (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Oral Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Allergy/Immunology (Other) (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Hemoglobin Decreased (Blood and lymphatic system disorders) | 6 (14) | 4 (9) | 4 (5)
Pain (General disorders) | 18 (21) | 7 (10) | 7 (7)
Urinary Incontinence (Renal and urinary disorders) | 3 (3) | 0 (0) | 0 (0)
Weight Loss (Metabolism and nutrition disorders) | 5 (7) | 0 (0) | 0 (0)
Vision Blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Joint Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Ear, Nose and Throat examination abnormal (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Glucose Intolerance (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0)
Hypertension (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Depression (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Bruising (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Fecal Incontinence (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Serum Magnesium Increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal Fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Weight Gain (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Extraocular Muscle Paresis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal (Other) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes